CLINICAL TRIAL: NCT00770393
Title: Randomized Phase III Trial Comparing Induction Chemotherapy Followed by Radiotherapy to Concomitant Chemoradiotherapy for Laryngeal Preservation in T3MO Pyriform Sinus Carcinoma
Brief Title: Laryngeal Preservation in Pyriform Sinus Carcinoma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Pr Jean-Michel PRADES, CHU de SAINT-ETIENNE
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0201089
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Last update posted 2008-10-10 (Estimated); Status verified 2008-10

CONDITIONS: Squamous Cell Carcinoma
Keywords: squamous cell carcinoma of the pyriform sinus; laryngeal preservation; patients with biopsy-proven previously untreated resectable T3 with fixed cord involvement squamous cell carcinoma of the pyriform sinus
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — Induction Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Cisplatin was administered intravenously at a dose of 100 mg/m2 on day 1 and fluorouracil was administered at a dose of 1 000 mg/m2/day by continuous intravenous infusion on day 1 to 5 for 2 courses after 3 weeks. After induction chemotherapy patients underwent ears, nose and throat examination and computed tomography imaging.
  Interventions: Procedure: induction chemotherapy
- 2 (Active Comparator): Intravenous cisplatin at dose of 100 mg/m2 on days 1, 22 and 43 was administered concomitantly with conventional radiotherapy to the primary tumor and to the neck lymph nodes according to the pathological findings of the pre-treatment neck dissection at a total dose of 70 Gy.
  Interventions: Procedure: Conventionnal chemotherapy

INTERVENTIONS:
Procedure: induction chemotherapy — Cisplatin was administered intravenously at a dose of 100 mg/m2 on day 1 and fluorouracil was administered at a dose of 1 000 mg/m2/day by continuous intravenous infusion on day 1 to 5 for 2 courses after 3 weeks. After induction chemotherapy patients underwent ears, nose and throat examination and computed tomography imaging. If a complete response (CR) or partial response (PR) of more than 80% is identified in the primary tumor, the patient was offered conventional radiotherapy as part of the protocol treatment. Radiotherapy was administered in 35 fractions of 2 Gy each over a 7 weeks period to the primary tumor (50 Gy) and the neck lymph nodes. The dose to the pathologically positive nodes was supplemented (20 Gy) at a total dose of 70 Gy. Doses and schedules of radiotherapy were identical in both treatment arms of the study.
  Arms: 1
Procedure: Conventionnal chemotherapy — Intravenous cisplatin at dose of 100 mg/m2 on days 1, 22 and 43 was administered concomitantly with conventional radiotherapy to the primary tumor and to the neck lymph nodes according to the pathological findings of the pre-treatment neck dissection at a total dose of 70 Gy.
  - Surgery was recommended to all patients who had a response less than 80%, stable disease or progressive disease in the primary tumor. If surgery was not feasible, the treatment choice was left up to the investigator's discretion.
  Arms: 2

SUMMARY:
Patients were eligible if they had biopsy proven, previously untreated T3 with fixed cord involvement squamous cell carcinoma of the pyriform sinus.

The study compare conventional radiotherapy with concurrent cisplatin to induction chemotherapy with cisplatin fluorouracil followed by conventional radiotherapy. The primary end point was the preservation of the larynx. The secondary end points included toxicity, causes of death and survival rates.

DETAILED DESCRIPTION:
Objectives: To compare conventional radiotherapy with concurrent cisplatin to induction chemotherapy with cisplatin fluorouracil followed by conventional radiotherapy. The primary end point was the preservation of the larynx. The secondary end points included toxicity, causes of death and survival rates.

Design: Multicenter prospective randomized phase III trial. Setting: Academic tertiary care center. Patients: Seventy one adult patients with biopsy-proven previously untreated resectable T3 with fixed cord involvement squamous cell carcinoma of the pyriform sinus.

Main Outcomes Measures: Patients were evaluated for toxic reactions, and organ preservation and survival rates. Statistical analysis of overall survival and event free survival was performed using the Kaplan Meier method.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible if they had biopsy proven, previously untreated T3 with fixed cord involvement squamous cell carcinoma of the pyriform sinus.

Patients also had to have a performance status (PS)< 1, and normal organ functions as defined by an absolute neutrophil count > 1500 cells/microl, platelet count > 100 000 cells/microl and a calculated creatinine clearance of more than 50 ml/min.

Exclusion Criteria:

* Patients with T1, T2 or T4 or M1 (metastatic disease) were ineligible.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2002-02; Primary Completion 2005-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The primary end point was to compare the two treatment arms to define the best schedule of preservation of an intact larynx. | 2 years

SECONDARY OUTCOMES:
Secondary end points analyzed causes of death, overall survival rate and event (loco-regional recurrent disease, metastases, death) free survival rate. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel PRADES, Pr, Principal Investigator — CHU de SAINT-ETIENNE
Locations (7):
- France (7):
  - CALLOC'H, Aix-les-Bains
  - LITAS, Le Puy
  - PIGNAT, Lyon
  - MAYAUD, Montbrison
  - Crampette, Montpellier
  - Lallemant, Nîmes
  - LACHEB, Roanne